CLINICAL TRIAL: NCT07026994
Title: Colchicine for the Prevention of Recurrence in Cerebral Amyloid Angiopathy RElated IntraCerebral Hemorrhage (CARE-ICH)
Brief Title: Colchicine for the Prevention of Recurrence in Cerebral Amyloid Angiopathy RElated IntraCerebral Hemorrhage
Acronym: CARE-ICH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Xin Cheng, Professor and Vice Chair, Department of Neurology, Huashan Hospital, Fudan University, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY2025-728
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Amyloid Angiopathy; Intracerebral Hemorrhage Lobar
Keywords: Cerebral Amyloid Angiopathy; Intracerebral Hemorrhage; Colchicine; Recurrence
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Cerebral Hemorrhage; Recurrence | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, phase II pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine group (Experimental): Patients in this arm will receiver oral colchicine 0.5mg once per day for 1 year combined with standard treatment
  Interventions: Drug: Colchicine 0.5mg
- Placebo group (Placebo Comparator): Patients in this arm will receiver oral matching placebo once per day for 1 year combined with standard treatment
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Colchicine 0.5mg — Oral colchicine 0.5mg once per day combined with standard treatment
  Arms: Colchicine group
Drug: Matching placebo — Oral matching placebo once per day combined with standard treatment
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to assess the safety and tolerability of colchicine for preventing intracerebral haemorrhage (ICH) recurrence in patients with cerebral amyloid angiopathy (CAA)-ICH at high risk of recurrence.

The main questions it aims to answer are:

* Is colchicine safe for CAA-ICH patients?
* Is colchicine well tolerated for CAA-ICH patients? Researchers will compare colchicine to a placebo (a look-alike substance that contains no drug) to see if colchicine is safe and tolerable for CAA-ICH patients and works to prevent ICH recurrence.

Participants will:

* Take colchicine or a placebo every day for 12 months
* Receive telephone follow-ups at 3 and 9 months, and visit the clinic at 6 and 12 months for checkups and tests
* Control blood pressure and improve lifestyle

DETAILED DESCRIPTION:
The CARE-ICH study is a multicenter, randomized, double-blind, placebo-controlled, phase II trial. The primary objective of the CARE-ICH study is to assess the safety and tolerability of colchicine for preventing ICH recurrence in patients with CAA-ICH at high risk of recurrence, as well as provide a preliminary estimate of the feasibility and efficacy for planning a phase III trial.

Patients with CAA-ICH and a high risk of recurrence-defined as 1 prior symptomatic ICH and presence of cortical superficial siderosis, or ≥2 prior symptomatic ICHs-within 3 months of their most recent ICH will be enrolled and randomized in a 1:1 ratio to receive either oral colchicine 0.5 mg once per day or matching placebo for 1 year, in addition to standard care, including blood pressure control and lifestyle modifications. Follow-up visits will take place at 3, 6, 9, and 12 months. Each visit will include assessments of adverse events, medication adherence, and clinical outcomes. The primary outcomes are the incidence of treatment-emergent adverse events and treatment tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥55 years;
* Diagnosed with "probable CAA with supporting pathology" or "probable CAA" according to the modified Boston criteria (version 1.5);
* High risk of recurrent ICH, defined as: 1 prior symptomatic ICH and presence of cortical superficial siderosis (cSS), or ≥2 prior symptomatic ICHs;
* Time interval since symptom onset of the most recent ICH: ≤3 months (earlier enrollment is preferred if criteria are met);
* Modified Rankin Scale (mRS) score ≤4 at randomization;
* Written informed consent from the participant or their legally authorized representative before study enrollment.

Exclusion Criteria:

* Secondary causes of ICH;
* Pre-existing moderate-to-severe renal, liver or blood disorders (anaemia [hemoglobin <10g/dL], thrombocytopaenia [platelet count <100×109/L], leucopenia [white blood cell <3×109/L], cirrhosis or severe hepatic dysfunction, renal insufficiency [estimated glomerular filtration rate (eGFR) <15mL/min]);
* Prior diagnosis of gout, peripheral neuropathy, myopathy, inflammatory bowel disease or chronic diarrhea;
* Concurrent treatment with regular immune-suppressant (corticosteroids, cyclophosphamide, azathioprine, mycophenolate mofetil, rituximab), moderate-to-strong CYP3A4 inhibitors (atazanavir, clarithromycin, darunavir/ritonavir, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, tipranavir/ritonavir) or P-glycoprotein inhibitors (cyclosporine, ranolazine);
* Known allergy, sensitivity or intolerance to colchicine;
* Contraindications or inability to complete brain MRI or susceptibility weighted imaging (SWI) scans;
* Pregnancy or breastfeeding;
* Recent participation in any other interventional study in the past 30 days before enrollment;
* Not expected to survive the follow-up period;
* Inability to adhere to study procedures;
* Any condition in which investigators believe that participating in this study may be harmful to the patient.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAE) | Any time within 1 year
  Incidence of treatment emergent adverse events (TEAE)
Frequency of participants who are adherence to medicine without permanent discontinuation due to TEAE until the end of follow-up. | 1 year
  Frequency of participants who are adherence to medicine without permanent discontinuation due to TEAE until the end of follow-up

SECONDARY OUTCOMES:
Safety-Treatment-related adverse events (TRAE) | Any time within 1 year
  An AE assessed as having a causal relationship to the study product, and be classified as definitely, probably or possibly related AEs
Safety-TEAE according to Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3 | Any time within 1 year
  TEAE according to Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3
Feasibility-Recruitment rate | 1 year
  The mean number of participants randomized per site per year
Feasibility-Retention rate | 1 year
  Randomized participants who completed 1-year follow-up
Clinical efficacy-Recurrent symptomatic spontaneous lobar ICH | Any time within 1 year
  A new non-traumatic lobar ICH lesion confirmed on SWI or CT with corresponding symptoms
Clinical efficacy-Composite of major adverse cardiovascular events (MACE) | Any time within 1 year
  Stroke (ischemic, hemorrhagic or undefined), myocardial infarction, revascularization procedure for coronary, carotid or peripheral arterial disease, and vascular death
Clinical efficacy-Any individual MACE | Any time within 1 year
  Stroke (ischemic, hemorrhagic or undefined), myocardial infarction, revascularization procedure for coronary, carotid or peripheral arterial disease, and vascular death
Clinical efficacy-Cognitive outcome | 1 year
  Cognitive function assessed by the Montreal Cognitive Assessment (MoCA) (The total score ranges from 0 to 30, with higher scores indicating better cognitive function)
Clinical efficacy-Functional outcome | 3-month, 6-month and 1-year
  Functional outcome assessed by the modified Rankin scale (mRS) [mRS score ranges from 0 (no symptom) to 6 (death) and higher score means worse functional outcome]
Clinical efficacy-Quality of life | 1 year
  Quality of life assessed by the EuroQol Five-Dimension Five-Level (EQ-5D-5L) questionnaire, which consists of two parts. The descriptive system evaluates health across five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on five levels of severity, where higher levels indicate more severe problems. The visual analogue scale is rated from 0 (worst imaginable health state) to 100 (best imaginable health state), representing the patient's self-rated overall health.
Clinical efficacy-Blood inflammatory markers | 6 month and 1 year
  High-sensitivity C-reactive protein (hsCRP) and interleukin-6 (IL-6).
Radiological efficacy-New asymptomatic ICH lesion | 1 year
  A new hemorrhagic lesion confirmed on SWI at 1-year, which was absent on SWI at baseline and was not associated with any acute neurological deficit
Radiological efficacy-Severe cSS progression | 1 year
  ≥2 new cSS foci on 1-year SWI scan
Radiological efficacy-Any cSS progression | 1 year
  ≥1 new cSS foci on 1-year SWI scan
Radiological efficacy-CMB progression | 1 year
  ≥5 new CMBs on 1-year SWI scan

OTHER OUTCOMES:
Exploratory outcomes-Blood-brain barrier permeability | 1 year
  Water exchange rate (kw) measured by diffusion-prepared pseudocontinuous arterial spin labeling (DP-pCASL) imaging
Exploratory outcomes-Glymphatic function | 1 year
  The index for diffusivity along the perivascular space (ALPS index) measured by diffusion tensor imaging
Exploratory outcomes-Neuroinflammation pattern | 1 year
  The standardized uptake value ratio of 18F-DPA-714 measured by translocator protein (TSPO)-PET

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Huashan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study can be made available to other researchers on reasonable request and after signing appropriate data sharing agreements.